CLINICAL TRIAL: NCT01820416
Title: The Effect of Low-Level Laser Stimulation on Hearing Thresholds
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Analysis showed no clinically or statistically significant effects
Sponsor: University of Iowa (Other)
Collaborators: GN Resound (Other)
Responsible Party: Principal Investigator, Shawn Goodman, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 200808718
Record Dates: First submitted 2013-03-25; First posted 2013-03-28 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-04

CONDITIONS: Hearing Loss
Keywords: Hearing Loss, Bilateral; Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss; Hearing Loss, Bilateral; Hearing Loss, Sensorineural | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low-Level Laser Therapy (Experimental): Low-level laser applied for approximately 4 minutes to the area around the pinna, the back of the neck, and the top of the head.
  Interventions: Radiation: Low-level Laser Therapy
- Disabled Laser (Placebo Comparator): Low-level laser device with laser diodes disabled. Also applied for approximately 4 minutes to the area around the pinna, the back of the neck, and the top of the head.
  Interventions: Other: Placebo Comparator: Disabled Laser
- Control (No Intervention): Visit laboratory using same schedule as experiment and placebo. No Low-level laser or any treatment applied. Used to assess normal test-retest variability.

INTERVENTIONS:
Radiation: Low-level Laser Therapy — Portable unit containing two laser diodes producing 532 and 635 nm wavelengths. Both diodes produced energy levels of 7.5 mw (class IIIb). Beams from both diodes were dispersed through lenses to create parallel line-generated beams, rather than spots. The 532 nm light was constant, and the 635 nm light was pulsed, with frequencies of 15 and 33 Hz. The pulsing alternated between frequencies every 30 seconds.
  Other Names: Erchonia EHL laser (Erchonia Medical, Inc.)
  Arms: Low-Level Laser Therapy
Other: Placebo Comparator: Disabled Laser — Portable unit containing two DISABLED laser diodes. Same protocol was followed as for the Experimental (radiation) group, except that the disabled diodes produced no radiation.
  Arms: Disabled Laser

SUMMARY:
The purpose of this study is to determine whether low-level laser therapy can improve hearing thresholds in individuals with hearing loss. Subjects will be randomly assigned to a treatment, placebo, or control group. The treatment group will be given a three treatment of low-level laser therapy, which consists of shining low-level lasers beams onto the ear and head. The laser beams are cool to the touch, and do not cause discomfort. Each laser treatment will last approximately 4 minutes. Three treatments will be applied three times within the course of one week. Hearing tests will be administered immediately before treatment, immediately after treatment, and six weeks after treatment. Results will be analyzed to determine the effect of the laser treatment on hearing.

DETAILED DESCRIPTION:
Low-level laser therapy has been practiced for about 20 years in Europe and is beginning to be practiced in the US. Theoretically, laser energy in the red and near infrared light spectrum is capable of penetrating 2-5 cm into tissue and can stimulate mitochondria in the cells to produce more energy (through the production of adenosine triphosphate), which in turn may help prevent or repair tissue damage. The effects of low-level laser therapy on hearing have not been well studied. It has been suggested that laser therapy might help repair damage to the cochlea and restore some degree of hearing loss. Studies of low-level laser stimulation of cochleae utilizing microscopy, PET imaging, and MRI suggest potential therapeutic benefit to hearing. While preliminary studies suggest a possible improvement in hearing thresholds, a carefully controlled study is needed to verify the results using a valid battery of audiological tests.

ELIGIBILITY:
Inclusion Criteria:

* bilateral sensorineural hearing loss
* normal middle ear status

Exclusion Criteria:

* pregnant or lactating
* serious mental health illness or medical/psychiatric hospitalization
* treatment with cancer chemotherapeutic agents or aminoglycoside antibiotics
* taking Aspirin, Ibuprofen, Naprosyn, Aleve
* taking any Quinine-related drugs
* taking any loop diuretics
* have a developmental disability or cognitive impairment
* history of drug abuse
* involved in litigation or claim related to hearing loss
* regularly exposed to significant occupational or recreational noise
* have a photosensitivity disorder
* have a retinal disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shawn S Goodman, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Goodman SS, Bentler RA, Dittberner A, Mertes IB. The effect of low-level laser therapy on hearing. ISRN Otolaryngol. 2013 Apr 23;2013:916370. doi: 10.1155/2013/916370. eCollection 2013. PMID 24024040

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low-Level Laser Therapy | Disabled Laser | Control
Started | 12 | 12 | 11
Completed | 9 | 10 | 11
Not Completed | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-Level Laser Therapy | Disabled Laser | Control | Total
Number analyzed (Participants) | 12 | 12 | 11 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.33 (15.37) | 55.58 (11.42) | 47.09 (16.71) | 51.46 (14.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 5 | 16
  Male | 6 | 7 | 6 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 11 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change in Speech Perception
Description: Hearing status, as assessed by the Connected Sentence Test (CST). Difference scores (post-test - pretest) are reported. The CST approximates everyday conversation. Scoring is based on the number of correctly repeated key words. Higher numbers indicate better scores. The minimum score is 0 (0%) and the maximum is 100 (100%). When comparing test-retest scores for an individual, Cox et al. (1988) suggest that changes of 15% or more (based on 100 key words) are indicative of significant changes. We subtracted the post-test from the pre-test, so that negative difference scores indicate worse performance, and positive difference scores indicate better performance. Difference scores with an absolute value smaller than 15 are interpreted as no significant change. In addition, pre- and post-test performance was assessed for groups using t-tests on the difference scores.
Time Frame: 7-10 days after baseline measures recorded
Measure: Mean (Standard Deviation); unit: difference scores
Arm/Group | Low-Level Laser Therapy | Disabled Laser | Control
Number analyzed (Participants) | 9 | 10 | 11
difference scores | -1.571 (6.949) | 2.286 (8.46) | -2.8 (5.329)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the time that the study was being conducted (from 09/01/2009 to 12/31/2009).
Arm/Group | Low-Level Laser Therapy | Disabled Laser | Control
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No